CLINICAL TRIAL: NCT05214677
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of DW1809 and DW1809-1 in Healthy Adult Volunteers
Brief Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Characteristics of DW1809
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW1809-103
Record Dates: First submitted 2021-12-12; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Back Pain; Acute Upper Respiratory Tract Infection
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): cross-over
  Interventions: Drug: DW1809; Drug: DW1809-1
- Sequence B (Experimental): cross-over
  Interventions: Drug: DW1809; Drug: DW1809-1

INTERVENTIONS:
Drug: DW1809 — pelubiprofen 30mg
  Other Names: Test
Drug: DW1809-1 — pelubiprofen 30mg (PELUBI tab.)
  Other Names: Reference

SUMMARY:
Randomized, Open-label, Oral, Single-dose, two-Sequence, four-Period, crossover study

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers who are ≥19 years old
* Body weight ≥50.0 kg and BMI between 18.0 and 30.0 kg/m2 and

Exclusion Criteria:

* Clinically significant Medical History
* In the case of women, pregnant(Urine-HCG positive) or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-09-07 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | up to 8 hour
  Pharmacokinetics of Pelubiprofen
Area under the plasma concentration versus time curve (AUC) | up to 8 hour
  Pharmacokinetics of Pelubiprofen

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea